CLINICAL TRIAL: NCT02852239
Title: A Phase I, Open Label, Multicenter, Single Dose Study to Evaluate the Pharmacokinetics of Dabrafenib in Healthy Subjects With Normal Renal Function and Subjects With Impaired Renal Function
Brief Title: Pharmacokinetics of Dabrafenib in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CDRB436A2106
Record Dates: First submitted 2016-07-26; First posted 2016-08-02 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-07

CONDITIONS: Renal Impairment
Keywords: Renal impairment; Healthy volunteers; Clinical pharmacology study; DRB436; dabrafenib; normal renal function; impaired renal function
MeSH Terms: conditions — Renal Insufficiency | interventions — dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 - Normal renal function (Experimental): Subjects with normal renal function defined as GFR ≥ 90 mL/min at baseline and matching to the renal impaired subject based on gender, race, age, and weight.
  Interventions: Drug: dabrafenib
- Group 2 - Severe renal function (Experimental): Subjects with severe renal impairment defined as GFR of 15-29 mL/min at baseline.
  Interventions: Drug: dabrafenib
- Group 3 - End stage renal disease (ESRD) (Experimental): Subjects with end stage renal disease (ESRD), defined as GFR of <15 mL/min at baseline.
  Interventions: Drug: dabrafenib

INTERVENTIONS:
Drug: dabrafenib — Single dose dabrafenib 100 mg
  Other Names: DRB436

SUMMARY:
To characterize the pharmacokinetics and safety of dabrafenib following a single 100 mg oral dose in subjects with severe renal impairment and end stage renal disease not on dialysis.

DETAILED DESCRIPTION:
The main objective of this trial is to evaluate the pharmacokinetics of dabrafenib and metabolites after a single oral dose of dabrafenib in subjects with renal impairment as compared to healthy subjects with normal renal function.

This was a single-dose, open-label, parallel group single dose study to evaluate the pharmacokinetics (PK) and safety of a single oral dose of dabrafenib 100 mg in subjects with severe RI or ESRD compared to matched healthy subjects with normal renal function (control group).

The study consisted of a screening period, a treatment period and a follow-up period.

The Screening period started up to 28 days prior to dosing. Subjects who satisfied the inclusion/exclusion criteria at screening were admitted for baseline evaluations, which was done locally by the investigator. In the treatment period, subjects received a single 100 mg oral dose of dabrafenib administered as two 50 mg capsules with a whole glass of non-carbonated water (approximately 240 mL) in the morning of Day 1 following an overnight fast (minimum 10 hours). Subjects were confined to the study facility from Day -1 to Day 5, for collection of serial blood and urine samples. Subjects were discharged on Day 5.

In the follow-up period a telephone call was made to subjects 30 days post-dose to evaluate subject safety during the weeks after discharge from the facility. Adverse events occurring prior to Day 30 were followed until resolution or until judged to be permanent. Subjects returned to the clinic on Days 90 and 180 for the post-dose dermatological examination follow up.

For this study, the terms "investigational drug", "study drug" or "study treatment" refer to dabrafenib, administered as a single dose.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Females must be of non-childbearing potential or must have negative pregnancy results at screening
* Good health as determined by lack of clinically significant findings
* Subjects must have a BMI between 18.0 kg/m2 and 38.0 kg/m2, with a body weight of at least 50 kg and no more than 140 kg
* Vitals signs within normal range
* Laboratory values at screening within local normal ranges or considered non-clinically significant

Additional criteria for renal impairment subjects:

-Stable renal disease without evidence of renal progression in the past 28 days prior to dosing

Additional criteria for healthy matched subjects:

* Matched to at least 1 renal impairment subject by race, age (+/-10 years), gender and weight (+/-10%)
* An absolute GFR of at least 90 ml/min

Exclusion Criteria for all subjects:

* Significant acute illness within the two weeks prior to dosing
* History or current diagnosis of cardiac disease indicating significant risk such as uncontrolled or significant cardiac disease or clinically significant ECG abnormalities
* Subjects will be screened for drugs of abuse
* History of drug or alcohol abuse within 6 months prior to dosing or evidence of such abuse as indicated by laboratory values at screening or baseline.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs.
* History of malignancy of any organ system, treated or untreated, within 5 years, regardless of where there is recurrence or metastases.
* Use of drugs known to prolong the QT interval within 4 weeks prior to dosing and for the duration of the study.
* Use of drugs know to affect CYP3A4 and/or CYP2C8 including both (strong or moderate) inhibitors and inducers, within 7 days prior to dosing or during the current study are prohibited

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Predose through 96 hours postdose
  The maximum (peak) observed plasma drug concentration after a single dose of dabrafenib
Area under the curve (AUClast) | Predose through 96 hours postdose
  AUClast is the area under the curve calculated to the last quantifiable concentration point after a single dose of dabrafenib
Area under the curve (AUFinf) | Predose through 96 hours postdose
  AUCinf is the area under the plasma concentration time curve extrapolated to infinity after a single dose of dabrafenib
Systemic drug clearance (CL/F) | Predose through 96 hours postdose
  Systemic clearance from plasma of dabrafenib after a single dose
Time to reach maximum concentration (Tmax) | Predose through 96 hours postdose
  The time to reach maximum (peak) concentration of dabrafenib after a single dose
Terminal elimination rate (Lambda_z) | Predose through 96 hours postdose
  Terminal elimination rate of dabrafenib after a single dose
Elimination half-life (T1/2) | Predose through 96 hours postdose
  Elimination half-life of dabrafenib after a single dose
Volume of distribution (Vz/F) | Predose through 96 hours postdose
  The apparent volume of distribution during the terminal elimination phase of dabrafenib after a single dose
Unchanged drug excreted in urine (Aet) | Predose through 96 hours postdose
  The amount of unchanged dabrafenib excreted in urine after a single dose
Renal clearance (CLr) | Predose through 96 hours postdose
  Renal clearance of dabrafenib calculated using plasma AUC after a single dose

SECONDARY OUTCOMES:
Number of subjects with adverse events | Time of drug administration through 30 days postdose
  Assess the safety of a single dose of dabrafenib through AE reports of subjects from drug administration through 30 days postdose
Number of subjects with abnormal lab values related to study drug | Time of study drug administration through 30 days postdose
  Assess the safety of a single dose of dabrafenib through hematology and chemistry blood tests
Number of subjects with abnormal blood pressure related to study drug | Time of study drug administration through 30 days postdose
  Assess the safety of a single dose of dabrafenib by monitoring changes in blood pressure
Changes in electrocardiogram (ECG) | Time of study drug administration through 30 days postdose
  Assess the safety of a single dose of dabrafenib by monitoring changes in ECG
Number of subjects with abnormal pulse rate related to study drug | Time of study drug administration through 30 days postdose
  Assess the safety of a single dose of dabrafenib by monitoring changes in heart rate
Number of subjects with abnormal respiratory rate related to study drug | Time of study drug administration through 30 days postdose
  Assess the safety of a single dose of dabrafenib by monitoring changes in respiratory rate

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - Omega Research Consultants LLC, DeBary, Florida
  - Hassman Research Institute, Berlin, New Jersey
  - Wake Research Associates Oncology, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CDRB436A2106 sudy results on the Novartis results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17675